CLINICAL TRIAL: NCT00280007
Title: AVATACE-1: Bevacizumab (Avastin®) as Inhibitor of Collateral Tumor Vessel Growth During Transarterial Chemoembolisation (TACE) for Hepatocellular Carcinoma (HCC) a Pilot Trial
Brief Title: Transarterial Chemoembolisation Plus Bevacizumab for Treatment of Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety concerns in the treatment arm
Sponsor: Medical University of Vienna (Other)
Responsible Party: Markus Peck-Radosavljevic, M. D., Medizinische Universität Wien
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MPR-2
Record Dates: First submitted 2006-01-19; First posted 2006-01-20 (Estimated); Last update posted 2010-04-22 (Estimated); Status verified 2009-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; TACE; transarterial chemoembolisation; portal hypertension; angiogenesis; VEGF; bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hypertension, Portal | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): bevacizumab infusion evey 2 weeks
  Interventions: Drug: bevacizumab
- 2 (Placebo Comparator): placebo infusion
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab — bevacizumab 5 mg/kg i.v. every 14 days for 52 weeks
  Other Names: -avastin

SUMMARY:
Patients with liver cirrhosis and hepatocellular carcinoma will undergo transarterial chemoembolisation (TACE) as clinically indicated and will be randomized to receive bevacizumab or placebo every 2 weeks up to 1 year. Tumor response will be assessed using MR of the liver and PET-scanning.

It will be tested whether the addition of bevacizumab as angiogenic inhibitor will slow down tumor progression, reduce the need for re-embolisation and will improve patient survival.

DETAILED DESCRIPTION:
TACE is an established therapy for patients with advanced stage HCC not amenable to liver transplantation or resection and has been shown to significantly improve survival in these patients compared to no treatment (8). TACE takes advantage of the predominantly arterial blood supply of malignant liver tumors contrary to the surrounding normal liver tissue, which receives more blood supply through the portal venous system.

TACE leads to predictable tumor necrosis until new blood vessels grow into the tumor margins to support tumor growth. Quite often after cutting off the blood supply through the hepatic artery, the tumor induces active angiogenesis to promote collateral blood vessel growth from liver capsule arteries or collaterals from the gastroduodenal artery. VEGF seems to be an important player in inducing this angiogenetic activity and tumor control and survival of patients after TACE have been linked to serum VEGF-levels with higher levels showing reduced survival.

Inhibition of these neoangiogenetic activity could lead to significantly improved in tumor control and survival in patients with advanced stage HCC.

2. STUDY OBJECTIVE

* to assess the effectiveness of bevacizumab in combination with TACE as measured by patients without tumor progression on MRT after 3 cycles of TACE as well as the number of TACE cycles applied for recurrent tumor after a maximum of one year treatment with bevacizumab
* to assess collateral tumor vessel growth on MRT / CT

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed HCC not suitable for OLT or resection (>3 nodules, >5 cm diameter, vascular invasion, clinically significant portal hypertension, other contraindications against OLT) or patients awaiting OLT with an expected waiting time >12 months
* Child-Pugh Stage A and B
* Liver disease of any etiology
* Written informed consent (approved by the Institutional Review Board [IRB]/Independent Ethics Committee [IEC]) obtained prior to any study specific screening procedures
* Patient must be able to comply with the protocol
* Age ≥18 years
* Women of childbearing potential must have a negative serum pregnancy test done 1 week prior to the administration of the study drug. Fertile women and men of childbearing potential (<2 years after last menstruation in women) must use effective means of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile)
* Proteinuria at baseline:

  * Urine dipstick of proteinuria <2+. Patients discovered to have >2+ proteinuria on dipstick urinalysis at baseline, should undergo a 24-hour urine collection and must demonstrate less <= 1 g of protein/24 hr.
* Haematology:

  * Absolute neutrophil count (ANC) > 1 x 109/L
  * Platelet count > 40 x 109/L
  * Haemoglobin > 9 g/dL (may be transfused to maintain or exceed this level)
  * Prothrombin time >= 40%
* Biochemistry:

  * Total bilirubin <= 5 mg/dL
  * Serum creatinine < 3.0 mg/dL
  * Life expectancy of >3 months

Exclusion Criteria:

* extra hepatic tumor spread
* complete portal vein thrombosis (common trunk)
* Child-Pugh-Stage C
* Prior TACE or TAE
* Other experimental therapies for HCC
* Acute variceal bleeding within the last 2 weeks
* Large oesophageal varices (>5 mm diameter) without prophylactic band ligation
* Past or current history (within the last 2 years prior to randomisation) of malignancies except for the indication under this study and curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix
* History or evidence upon physical examination of CNS disease unless adequately treated (e.g., seizure not controlled with standard medical therapy or history of stroke within < 6 months), excluding hepatic encephalopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study
* Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants for therapeutic purposes
* Chronic, daily treatment with aspirin (>325mg/day)
* Pregnancy (positive serum pregnancy test) or lactation
* Uncontrolled hypertension
* Serious, non-healing wound, ulcer, or bone fracture
* Patients with known allergy to Chinese hamster ovary cell proteins or other recombinant human or humanized antibodies or to any excipients of Bevacizumab formulation; or to any other study drugs
* Currently or recent (within the 30 days prior to starting study treatment) treatment of another investigational drug or participation in another investigational study
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤ 6 months prior to randomisation), myocardial infarction (≤ 6 months prior to randomisation), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication
* Evidence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or patient at high risk from treatment complications

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
to assess the effectiveness of bevacizumab in combination with TACE as measured by patients without tumor progression after a maximum of one year treatment with bevacizumab | 12 months
to assess collateral tumor vessel growth on MRT / CT after 3, 6, and 12 months | 12 months

SECONDARY OUTCOMES:
overall survival | 12 months
time to progression | 12 months
safety | 12 months
total number of TACE-cycles applied | 12 months
metabolically active tumor size on PET-scan | 12 months
circulating endothelial progenitors and pro-angiogenic hematopoietic cells as markers of angiogenesis | 12 months
HGF-levels during therapy | 12 months
portal hypertension and systemic hemodynamics | 12 months
cost | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Markus Peck-Radosavljevic, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medizinische Universität Wien, Vienna, Austria